CLINICAL TRIAL: NCT05414682
Title: Brain Healthy Soul Food Diet Intervention Among Older African Americans (Aim 2-3)
Brief Title: Brain Healthy Soul Food Diet Intervention Among Older African Americans
Acronym: MIND+SOUL Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 148307
Record Dates: First submitted 2022-05-19; First posted 2022-06-10 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases; Cognitive Decline
MeSH Terms: conditions — Cardiovascular Diseases; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIND+SOUL Diet (Experimental): The MIND+SOUL diet is an adapted brain-healthy soul food diet. Participants follow the diet for 12 weeks.
  Interventions: Other: MIND+SOUL Diet

INTERVENTIONS:
Other: MIND+SOUL Diet — The MIND+SOUL Diet is an adapted brain-healthy soul food diet.

SUMMARY:
The primary goal of this project is to evaluate feasibility and acceptability of the MIND+SOUL diet and its implementation. Secondary goals of this project are to evaluate cardiovascular risk profile, nutritional health status, and cognition in relation to the MIND+SOUL diet intervention.

DETAILED DESCRIPTION:
This is a single arm trial designed to pilot test an adapted brain healthy diet intervention among older AA (n=30). Specifically, this study aims to evaluate the feasibility and acceptability of the brain healthy soul food diet intervention. As secondary outcomes, this study aims to assess body composition, cardiovascular risk, nutritional health status, and changes in cognition among older AA to form the basis of estimating power and sample size for a future full-scale randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American or Black
* Age 55 and older
* English Proficient
* 1 or more of the following CVD risk factors (high blood pressure, high cholesterol, overweight/obesity with a BMI of 25 or more)
* Cognitively Normal with an AD8 <2 (normal cognition)

Exclusion Criteria:

* No CVD risk factors
* AD8 equal to or greater than 2
* Existing diet plan prescribed by a clinician
* Non menopausal (because of DXA scan)
* No internet connection
* Uncontrolled hypertension, by history, or as indicated by supine systolic blood pressure >165 mmHg or diastolic blood pressure >95 mmHg at the baseline visit. If an initial blood pressure reading is higher than this, an additional attempt (at this visit or on another day) could be used before excluding a patient for uncontrolled hypertension
* Neurological diseases that impact cognition
* Other medical conditions likely to be negatively impacted by a diet change or that could confound the study data
* Unable or unwilling to provide written consent
* PI determination that study is unsafe or unsuitable
* Active depression as determined by a score of 5 or above on the PHQ9 and deemed to be clinically significant by the medical monitor

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaw AR, Honea R, Mudaranthakam DP, Young K, Vidoni ED, Morris JK, Billinger S, Key MN, Berkley-Patton J, Burns JM. Feasibility of the MIND+SOUL Culturally Tailored Brain Healthy Diet: A Pilot Study. Am J Lifestyle Med. 2024 Oct 23:15598276241296052. doi: 10.1177/15598276241296052. Online ahead of print. PMID 39540187

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MIND+SOUL Diet
Started | 29
Completed | 25
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (6.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Cardiovascular Risk Factor [Count of Participants; unit: Participants]
  high blood pressure | 29
  high cholesterol | 29
  overweight (BMI greater or equal to 25) | 29
Cognitively Normal [Count of Participants; unit: Participants] | 29
No active depression [Count of Participants; unit: Participants] | 29

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Retention Rate
Description: Feasibility will be assessed by retention rate. This will be calculated as the percentage of participants who complete all aspects of the intervention including cooking classes and coach directed dietary call support.
Time Frame: 12 weeks
Population: All participants who enrolled in the MIND+SOUL pilot and completed baseline assessments were included in the feasibility analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
percentage of participants | 28 [14.3 to 47.6]

2. Secondary Outcome: Total Fat Mass
Description: Total fat mass was assessed using dual-energy X-ray absorptiometry (DXA) to measure total fat mass. Assessments were conducted at baseline and again at the 12-week follow-up. The values reported below reflect the 12-week follow-up, with changes calculated from baseline to 12 weeks.
Time Frame: Assessed at baseline and 12 weeks; 12-week data reported
Population: Participants who completed both baseline and 12-week DXA body composition assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
grams | 37,395.1 (13,218.4)

3. Secondary Outcome: Android Fat Mass
Description: Android fat mass was assessed using dual-energy X-ray absorptiometry (DXA) to measure android fat mass. Assessments were conducted at baseline and again at the 12-week follow-up. The values reported below reflect the 12-week follow-up, with changes calculated from baseline to 12 weeks.
Time Frame: Assessed at baseline and 12 weeks; 12-week data reported
Population: Participants who completed both baseline and 12-week DXA body composition assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
grams | 3,301.2 (1,749.3)

4. Secondary Outcome: Waist Circumference
Description: Waist circumference was measured using a standard tape measure at baseline and 12 weeks. Data reported reflect 12-week follow-up values for participants who completed both time points.
Time Frame: Assessed at baseline and 12 weeks; 12-week data reported
Population: Participants who completed both baseline and 12-week DXA body composition assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
cm | 98.5 (14.0)

5. Secondary Outcome: Body Mass Index
Description: Body mass index was calculated using measured height and weight at baseline and 12 weeks. The value below reflects BMI at the 12-week follow-up for participants who completed both assessments.
Time Frame: Assessed at baseline and 12 weeks; 12-week data reported
Population: Participants who completed both baseline and 12-week DXA body composition assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
kg/m^2 | 34.6 (7.9)

6. Secondary Outcome: Total Cholesterol
Description: Cardiovascular risk profile will be measured by cholesterol. Cholesterol will be measured using the PTS Diagnostics Cardiocheck Plus Analyzer Cholesterol and Glucose Check.
Time Frame: All cardiovascular risk prolife assessments will be collected at baseline and at the 12-week mark.
Population: Participants who completed both baseline and 12-week assessments for cholesterol were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
mg/dL
  Cholesterol at baseline | 177.5 (36.46)
  Cholesterol at 12-weeks | 181.5 (53.88)

7. Secondary Outcome: Systolic Blood Pressure
Description: Cardiovascular risk profile will be measured by systolic blood pressure. Blood pressure will be measured using the Omron 5 series blood pressure monitor. C
Time Frame: All cardiovascular risk prolife assessments will be collected at baseline and at the 12-week mark.
Population: Participants who completed both baseline and 12-week assessments for blood pressure were included in this analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 29
mmHg
  Systolic blood pressure at baseline | 127.31 (12.421)
  Systolic blood pressure at 12 weeks | 132.40 (14.602)

8. Secondary Outcome: Skin Carotenoid Score (Veggie Meter) Skin Carotenoid Score (Veggie Meter) Skin Carotenoid Score (Veggie Meter)
Description: Skin carotenoid levels were assessed using the Veggie Meter®, which uses reflection spectroscopy to provide an objective measure of carotenoid-rich fruit and vegetable intake. Scores typically range from 0 to 800. Higher scores indicate higher carotenoid levels and greater intake of fruits and vegetables. Changes were evaluated from baseline to 12 weeks.
Time Frame: Self-reported dietary intake was assessed at baseline and at the 12-week follow-up.
Population: Participants who completed Veggie Meter assessments at both baseline and 12-week follow-up were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
score on a scale
  Skin Carotenoid Score (Veggie Meter) at baseline | 245.2 (96.45)
  Skin Carotenoid Score (Veggie Meter) at 12 weeks | 270.9 (91.24)

9. Secondary Outcome: Self-Reported Fruit and Vegetable Intake (NHANES Dietary Screener)
Description: Self-reported fruit and vegetable intake was assessed using the NHANES Dietary Screener Questionnaire (DSQ). The DSQ estimates average daily intake in cups per day, based on participant-reported consumption over the past 30 days. There is no fixed score range; higher estimated intake reflects greater fruit and vegetable consumption and better nutritional health. Changes were assessed from baseline to 12 weeks.
Time Frame: Self-reported dietary intake was assessed at baseline and at the 12-week follow-up
Population: Participants who completed the NHANES Dietary Screener at both baseline and 12-week follow-up were included in the analysis.
Measure: Mean (Standard Deviation); unit: cups per day
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
cups per day
  Self-Reported Fruit and Vegetable Intake (NHANES Dietary Screener) at baseline | 0.626 (0.5634)
  Self-Reported Fruit and Vegetable Intake (NHANES Dietary Screener) at 12 weeks | 0.891 (0.6052)

10. Secondary Outcome: Cognitive Function
Description: Cognitive function was assessed using the NIH Toolbox Cognition Battery. The following assessments were administered to evaluate specific cognitive domains: NIH Toolbox List Sorting Working Memory Test (working memory), Picture Vocabulary Test (language), Oral Reading Recognition Test (reading), Pattern Comparison Processing Speed Test (processing speed), and Flanker Inhibitory Control and Attention Test (executive function). Each test yields a fully normed T-score ranging from 0 to 200, with a normative mean of 100 and a standard deviation of 15. Higher scores reflect better cognitive performance. This outcome specifically focuses on changes in executive function, as measured by the Flanker Inhibitory Control and Attention Test. Scores were collected at two time points: baseline and 12 weeks. The value reported in the data table reflects the mean score at 12 weeks.
Time Frame: Cognitive function was assessed at baseline and again at 12 weeks. The data table reports the outcome value from the 12-week time point.
Population: Participants who completed NIH Toolbox cognitive assessments at both baseline and 12-week follow-up were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale from 0 to 200
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
Scores on a scale from 0 to 200 | 90.2 (4.1)

11. Secondary Outcome: Feasibility: Reasons for Refusal
Description: Feasibility was planned to be assessed by tracking reasons for refusal to participate during the recruitment phase. Staff aimed to document participant-reported reasons for non-enrollment during initial outreach and screening efforts, however staff did not document participant-reported reasons for non-enrollment.
Time Frame: Reasons for refusal were supposed to be tracked throughout the recruitment period, which lasted approximately three months, but were not tracked.
Population: No data is available for this outcome. The primary investigator did not build the database to include recording of participant-reported reasons for for non-enrollment, therefore the data was not collected.
Groups:
- MIND+SOUL Diet MIND+SOUL Diet MIND+SOUL Diet MIND+SOUL Diet MIND+SOUL Diet: The MIND+SOUL diet is a 12-week culturally tailored brain-healthy dietary intervention that includes group education, cooking classes, spiritual wellness resources, health coaching, and weekly groceries.
Arm/Group | MIND+SOUL Diet MIND+SOUL Diet MIND+SOUL Diet MIND+SOUL Diet MIND+SOUL Diet
Number analyzed (Participants) | 0

12. Secondary Outcome: Satisfaction - Visual Analog Scale
Description: Satisfaction with the MIND+SOUL diet was assessed using a Visual Analog Scale (VAS) for overall program satisfaction. The Visual Analog Scale is a single-item self-report tool ranging from 0 to 10, where 0 indicates the least amount of satisfaction and 10 indicates the highest level of satisfaction. Higher scores represent better outcomes, meaning greater satisfaction with the intervention.
Time Frame: Satisfaction assessment will be conducted at the 12-week mark.
Population: Participants who completed the Visual Analog Scale for satisfaction at the 12-week follow-up were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
Score on a scale | 9.4 (1.2)

13. Secondary Outcome: Acceptability
Description: Acceptability of the MIND+SOUL intervention was assessed using a REDCap-administered online survey developed to evaluate participant perceptions across five domains: affective attitude, burden, ethicality, perceived effectiveness, and self-efficacy. The survey includes 20 items, each scored on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 20 to 100, with higher scores indicating greater acceptability of the intervention. Scores were collected at the 12-week follow-up.
Time Frame: Acceptability assessment will be conducted at the 12-week mark.
Population: Participants who completed the post-intervention acceptability survey at the 12-week follow-up were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | MIND+SOUL Diet
Number analyzed (Participants) | 25
Score on scale | 91.8 (11.4)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the 12-week intervention period for each participant.
Description: Adverse events were monitored informally during routine check-ins across the 12-week intervention period. One participant reported feeling dehydrated, which they attributed to not having consumed water throughout the day. Another participant reported feeling bloated after consuming foods included in the study diet. These events were recorded during check-ins and monitored by study staff.
Arm/Group | MIND+SOUL Diet
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 2/29
OTHER ADVERSE EVENTS (reported when occurring in more than 0.08% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIND+SOUL Diet (N=29)
Dehydration (Gastrointestinal disorders) | 1 (1) — Dehydration
Bloating (Metabolism and nutrition disorders) | 1 (1) — Bloating

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT05414682/Prot_SAP_000.pdf